CLINICAL TRIAL: NCT03644641
Title: The Influence of Prone Position for Spinal Surgery on Visual Acuity, a Comparison of Volatile Anesthesia With Desflurane to Total Intravenous Anesthesia With Propofol
Brief Title: The Influence of Prone Position for Spinal Surgery on Visual Acuity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Principal Investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHospital Hradec Kral
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Vision; Disorder, Loss
Keywords: Desflurane; Near-infrared spectroscopy; Propofol; Spinal surgery; Prone position; Visual acuity; Visual loss
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane Group (Experimental): Induction and anesthesia will be held by using desflurane
  Interventions: Procedure: Desflurane Group
- Propofol Group (Experimental): Induction and anesthesia will be held by using target-control anesthesia with propofol
  Interventions: Procedure: Propofol Group

INTERVENTIONS:
Procedure: Desflurane Group — General anesthesia will be held using desflurane in end- tidal concentration according to target value of entropy levels (between 40 and 60).
  Arms: Desflurane Group
Procedure: Propofol Group — General anesthesia will be held using Schnider effect model for propofol (target control anesthesia). Titration will be done according to target value of entropy levels (between 40 and 60).
  Arms: Propofol Group

SUMMARY:
This study investigated the effect of desflurane and propofol anesthesia on visual acuity in patients in prone position for spinal surgery. Many trials have investigated the effects of different anesthetic agents on intraocular pressure, propofol may reduce intraocular pressure more than other intravenous anesthetics.

DETAILED DESCRIPTION:
Perioperative increase in intraocular pressure can be caused by prone positioning. In addition to surgical factors, patients with glaucoma, uncontrolled hypertension, arthrosclerosis, and morbid obesity are at risk for potentially damaging optic nerve and loss of optic nerve function. Some studies found that intraocular pressure values were significantly lower in patients undergoing propofol total intravenous anesthesia than in patients undergoing desflurane anesthesia during intraoperative positional changes. Pronounced vasodilatation caused by desflurane might produced hyperaemia with higher intraocular pressure. Hemodynamic response to prone position measured by near-infrared spectroscopy (NIRS) on the prefrontal cortex could determine changes caused by prone position.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma scale 15
* American Society of Anesthesiologists (ASA) Physical Status Classification System I-III
* spinal surgery in duration less than 3 hours
* sinus rhythm

Exclusion Criteria:

* postoperative artificial ventilation
* serious neurological disease
* lung disease with hypercapnia
* propofol allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual injury | 48 hours
  worsening of test for visual acuity (Rodenstock)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Dostal, MD, Ph.D., Study Director — Hradec Kralove, Czechia 50005
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia